CLINICAL TRIAL: NCT02527733
Title: Retinal Sensitivity in Branch Retinal Vein Occlusion After Anti-VEGF Therapy
Brief Title: Retinal Sensitivity in BRVO After Anti-VEGF Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fukushima Medical University (Other)
Responsible Party: Principal Investigator, Akira Ojima, Assistant Professor, Fukushima Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2129
Record Dates: First submitted 2015-06-29; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab; Lasers

ARMS (2):
- Ranibizumab (Active Comparator): After initial single intravitreal injection of ranibizumab (0.5mg), participants receive monthly as-needed injection of ranibizumab (0.5mg) when visual acuity is less than 1.0 and foveal thickness is more than 250 micrometers.
  Interventions: Drug: Ranibizumab
- Ranibizumab and laser (Active Comparator): After initial single intravitreal injection of ranibizumab (0.5mg), participants receive monthly as-needed injection of ranibizumab (0.5mg) when visual acuity is less than 1.0 and foveal thickness is more than 250 micrometers. Macular laser photocoagulation will be performed when visual acuity is less than 1.0 and foveal thickness is more than 250 micrometers.
  Interventions: Drug: Ranibizumab and laser

INTERVENTIONS:
Drug: Ranibizumab
  Arms: Ranibizumab
Drug: Ranibizumab and laser
  Arms: Ranibizumab and laser

SUMMARY:
The efficacy of anti-vascular endothelial growth factor (VEGF) therapy for branch retinal vein occlusion (BRVO) is shown, but its effect on retinal sensitivity is not fully investigated. The purpose of this study is to compare the changes in retinal sensitivity after ranibizumab therapy or combination therapy of ranibizumab and laser photocoagulation in eyes with BRVO.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive patients of branch retinal vein occlusion with visual acuity of less than 1.0 and macular edema of more than 250 micrometers in foveal thickness.

Exclusion Criteria:

* Patients with history of treatment for branch retinal vein occlusion, possibility of pregnancy, allergy for ranibizumab, intraocular infection, or severe inflammation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Retinal sensitivity measured by microperimetry (MP-3, NIDEK, Japan) | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Fukushima Medical University, Fukushima, Fukushima, Japan